CLINICAL TRIAL: NCT04562142
Title: Validation of the CAD-det System, a Novel Non-Invasive Acoustic Diagnostic for the Diagnosis of Coronary Artery Disease (The CAD-det Validation Study)
Brief Title: A Novel Non-Invasive Acoustic Diagnostic for the Diagnosis of Coronary Artery Disease The CAD-det Validation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AusculSciences Canada Inc. (Industry)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAD-det Validation
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Atherosclerosis; Coronary Occlusion
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Atherosclerosis; Coronary Occlusion

STUDY DESIGN:
Intervention Model Description: CAD-det
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CAD-det — CAD-det test will be done on participants with suspected CAD clinically referred for ICA at a participating clinical investigation site.

SUMMARY:
The purpose of the study is to collect acoustic, ECG, and clinical data from consenting participants, so that AusculSciences can perform analysis on the sounds produced by the heart and determine the accuracy of the CAD-det System for detecting CAD.

DETAILED DESCRIPTION:
This is a prospective multi-center clinical trial. Using the CAD-det, acoustic and electrical cardiac data will be collected from participants with intermediate pretest probability of CAD who are referred to invasive coronary angiography (ICA). The CAD-det recording will be administered prior to the scheduled ICA procedure. The data collected by CAD-det will be processed using AusculSciences' Data Analysis Application (DAA) to produce a patient's indication for CAD.

ELIGIBILITY:
Inclusion Criteria:

1. Stable
2. >/= 19 years old
3. Suspected obstructive CAD
4. Referred to ICA

Exclusion Criteria:

1. Documented CAD or coronary revascularization
2. Age < 19 years old
3. Acute coronary syndromes
4. Congenital heart disease or heart transplantation
5. Dextrocardia
6. Uncontrolled irregular heart rhythm (atrial arrhythmia (fibrillation, flutter) or frequent PACs or PVCs (>10/minute))
7. Resting heart rate > 110 bpm
8. Known hemodynamically-significant valvular heart disease, audible diastolic murmurs, or hypertrophic or non-ischemic cardiomyopathy
9. Chest wall deformity or wounds in adhesive application areas
10. Pregnancy
11. Unwillingness or inability to provide informed consent or to comply with the study protocol

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
CAD-det to validate: | up to 1 Year
  CAD-det to detect obstructive CAD as defined as QCA diameter stenosis greater than or equal to 50%.

SECONDARY OUTCOMES:
CAD-det to detect: | up to 1 year
  1. Obstructive CAD as defined as QCA diameter stenosis greater than or equal to 50% stratified according to sex (men and women).
  2. Severity of CAD by QCA:
     1. 0 - 25% diameter stenosis (Negative for obstructive CAD);
     2. 25 - 50% diameter stenosis (Negative for obstructive CAD);
     3. 50 - 69% diameter stenosis (Positive for obstructive CAD);
     4. 70% or greater diameter stenosis (Positive for obstructive CAD); and
     5. Equivocal or non-diagnostic.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chow, MD, Principal Investigator — Ottawa Heart Institue Research Foundation
Locations (2):
- Canada (2):
  - The University of Ottawa Heart Institute, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makaryus AN, Makaryus JN, Figgatt A, Mulholland D, Kushner H, Semmlow JL, Mieres J, Taylor AJ. Utility of an advanced digital electronic stethoscope in the diagnosis of coronary artery disease compared with coronary computed tomographic angiography. Am J Cardiol. 2013 Mar 15;111(6):786-92. doi: 10.1016/j.amjcard.2012.11.039. Epub 2013 Jan 1. PMID 23290309
- See also: Study Sponsor — http://ausculsciences.com